CLINICAL TRIAL: NCT07403201
Title: The Effect of Combination Therapy Dlbs 3233 and Clomifen Citrate vs Clomifen Citrate on Homa ir, Maturation Follicle, and Menstrual Cycle in PCOS Cases at Muhammadiyah Asri Medical Center Hospital
Brief Title: The Effect of Therapy Combination in PCOS With Dlbs 3233
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Inlacinpenelitian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inlacinpenelitian
Record Dates: First submitted 2021-11-24; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: pcos; dlbbs 3233; clomifen citrat
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interprofessional collaboration treatment for PCOS at RS AMC Yogyakarta (No Intervention): to know the effect of interproffessional collaboration in pcos patient. And also to try give the best treatment for pcos patient
- The effectiveness Inlacin therapy vs clomiphene citrat to optimize AMH in PCOS (Experimental): To compare the effectiveness of treatment for women with pcos syndrome between inlacin and clomiphene citrat with knowing the AMH first
  Interventions: Combination Product: dlbs 3233 , clomifen citrat

INTERVENTIONS:
Combination Product: dlbs 3233 , clomifen citrat — combination theraphy
  Arms: The effectiveness Inlacin therapy vs clomiphene citrat to optimize AMH in PCOS

SUMMARY:
The effect of combination therapy dlbs 3233 and clomifen citrate vs clomifen citrate on homa ir, maturation follicle, and menstrual cycle in PCOS cases at Muhammadiyah Asri Medical Center Hospital

DETAILED DESCRIPTION:
to know the effect of combination dlbs 3233 theraphy and clomifen citrat in cases PCOS to control menstrual cycle and weight loss

ELIGIBILITY:
Inclusion Criteria:

* married agree to join this research

Exclusion Criteria:

* dis agree to join research

Max Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — women
Enrollment: 90 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-01-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in HOMA-IR | Baseline (Day 3 of menses) to 3 months (Day 3 of menses after treatment)
  HOMA-IR will be used to assess insulin resistance. Fasting glucose and fasting insulin will be collected on Day 3 of menses at baseline (pre-treatment) and after 3 months of treatment, and HOMA-IR will be calculated as a single index value.
Change in serum AMH concentration | Baseline (Day 3 of menses) to 3 months (Day 3 of menses after treatment)
  Serum anti-mullerian hormone (AMH) will be measured from venous blood collected on Day 3 of menses at baseline (pre-treatment) and after 3 months of treatment to assess ovarian function response.

SECONDARY OUTCOMES:
Change in total follicle count on Day 12 ultrasound | Baseline cycle (Day 12) to Month 3 cycle (Day 12)
  Total number of follicles will be assessed by transvaginal ultrasound on Day 12 of the menstrual cycle at baseline and after 3 months of treatment.
Change in number of mature follicles on Day 12 ultrasound | Baseline cycle (Day 12) to Month 3 cycle (Day 12)
  Number of mature follicles assessed by transvaginal ultrasound on Day 12 of the menstrual cycle at baseline and after 3 months of treatment.
Change in mature follicle diameter on Day 12 ultrasound | Baseline cycle (Day 12) to Month 3 cycle (Day 12)
  Mature (dominant) follicle diameter will be measured by transvaginal ultrasound on Day 12 of the menstrual cycle at baseline and after 3 months of treatment.
Menstrual cycle regularity during the 3-month treatment period | During the 3-month treatment period
  Proportion of participants who experience monthly menstrual bleeding during the 3-month treatment period.

OTHER OUTCOMES:
Change in body mass index (BMI) during treatment | Baseline to 3 months
  BMI calculated using measured weight and height at baseline and at the end of the 3-month treatment period.
Change in ovarian volume on ultrasound during annual follow-up | Up to 5 years (annual follow-up)
  Ovarian volume measured by transvaginal ultrasound at each annual follow-up visit after completion of the 3-month treatment period. Ovarian volume recorded as a numeric value (cm³).
Change in BMI during annual follow-up | Up to 5 years (annual follow-up)
  BMI calculated at each annual follow-up visit after completion of the 3-month treatment period using measured weight and height.

CONTACTS AND LOCATIONS:
Overall Officials: UMY Yogyakarta, Study Director — muhammadiyah university of yogyakarta
Locations (1):
- RS AMC Yogyakarta, Yogyakarta, DIY, Indonesia

IPD SHARING:
Plan to Share IPD: No